CLINICAL TRIAL: NCT07130175
Title: Efficacy of Radiofrequency Catheter Ablation on Improving Cardiac Function in Patients With Polymorphic Ventricular Tachycardia and Coexisting Heart Failure: A Randomized Controlled Trial
Brief Title: Radiofrequency Ablation for Polymorphic Ventricular Tachycardia With Heart Failure (RFCA for PMVT-HF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qian Feng (Other)
Collaborators: The First Hospital of Zhangjiakou City (Unknown)
Responsible Party: Sponsor-Investigator, Qian Feng, Principal investigator, The Second Affiliated Hospital of Hebei North University
Organization: The Second Affiliated Hospital of Hebei North University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022109
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Polymorphic Ventricular Tachycardia; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Radiofrequency Catheter Ablation (RFCA) Group (Experimental): Patients received Radiofrequency Catheter Ablation (RFCA) in addition to standard Guideline-Directed Medical Therapy (GDMT). GDMT included spironolactone 20 mg/day, metoprolol succinate 25 mg twice daily, and sacubitril/valsartan 50 mg twice daily, titrated as tolerated. Patients were followed for 6 months post-procedure.
  Interventions: Device: Radiofrequency Catheter Ablation; Drug: Guideline-Directed Medical Therapy (GDMT)
- Active Comparator: Control Group (Active Comparator): Patients received standard Guideline-Directed Medical Therapy (GDMT) alone. The regimen included spironolactone 20 mg/day, metoprolol succinate 25 mg twice daily, and sacubitril/valsartan 50 mg twice daily, titrated as tolerated. Patients were followed for 6 months.
  Interventions: Drug: Guideline-Directed Medical Therapy (GDMT)

INTERVENTIONS:
Device: Radiofrequency Catheter Ablation — An invasive procedure performed under local anesthesia. An electroanatomic mapping system (CARTO 3) was used to identify the arrhythmogenic substrate of the PMVT. Radiofrequency energy was delivered via an irrigated-tip catheter (30-35 W, 43°C, 17 mL/min saline irrigation) to ablate the target sites. The procedural endpoint was the non-inducibility of the clinical arrhythmia. Post-procedure, patients were prescribed amiodarone.
  Arms: Experimental: Radiofrequency Catheter Ablation (RFCA) Group
Drug: Guideline-Directed Medical Therapy (GDMT) — Standard medical therapy for heart failure, including spironolactone (20 mg once daily), metoprolol succinate (25 mg twice daily), and sacubitril/valsartan (50 mg twice daily). Doses were titrated according to patient tolerance and clinical guidelines.

SUMMARY:
This is a prospective, randomized, controlled trial to investigate the efficacy of radiofrequency catheter ablation (RFCA) combined with guideline-directed medical therapy (GDMT) compared to GDMT alone in patients with polymorphic ventricular tachycardia (PMVT) and coexisting heart failure (HF). The study aims to evaluate whether the addition of RFCA can lead to superior improvements in cardiac function, clinical outcomes, and serum biomarkers at a 6-month follow-up.

DETAILED DESCRIPTION:
The co-occurrence of polymorphic ventricular tachycardia (PMVT) and heart failure (HF) presents a significant clinical challenge with poor prognosis. While guideline-directed medical therapy (GDMT) is standard care, it may not adequately address the arrhythmic substrate. Radiofrequency catheter ablation (RFCA) has proven effective for other arrhythmias in the context of HF, but its role in PMVT is less established. This study tests the hypothesis that RFCA, as an adjunct to GDMT, is superior to GDMT alone in this high-risk population. A total of 118 eligible patients with PMVT and HF were randomized in a 1:1 ratio to receive either RFCA plus GDMT (Study Group) or GDMT alone (Control Group). The primary objective is to compare changes in cardiac function parameters (LVEF, LVEDV, LVESV, SV) assessed by Cardiac Magnetic Resonance (CMR) from baseline to 6 months post-treatment. Secondary objectives include evaluating differences in clinical efficacy, serum biomarkers of myocardial injury and fibrosis (H-FABP, sST2, Gal-3, TIMP-1), and the incidence of adverse events between the two groups. The findings aim to provide robust evidence for RFCA as a therapeutic strategy to improve cardiac function and clinical outcomes for patients with PMVT and HF.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of polymorphic ventricular tachycardia (PMVT) and coexisting heart failure (HF) via ECG and clinical evaluation.
* New York Heart Association (NYHA) functional class II-IV.
* First-time candidate for RFCA.
* Provided written informed consent.

Exclusion Criteria:

* Diagnosis of a malignant tumor.
* Severe psychiatric disorders.
* History of thyroid diseases or collagen diseases.
* Recent infectious diseases.
* Severe dysfunction of the lungs, liver, or kidneys.
* Coexisting coagulation disorders.
* Contraindications to amiodarone.
* Pregnancy or lactation.
* Congenital heart disease, cor pulmonale, or other primary structural heart diseases.
* Prior pacemaker implantation.
* Cardiac surgery within the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2022-12-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) | Baseline, 6 Months Post-treatment
  Measured by Cardiac Magnetic Resonance (CMR) imaging to assess global systolic function.
Change in Left Ventricular End-Diastolic Volume (LVEDV) | Baseline, 6 Months Post-treatment
  Measured by CMR to assess cardiac size and remodeling.
Change in Left Ventricular End-Systolic Volume (LVESV) | Baseline, 6 Months Post-treatment
  Measured by CMR to assess cardiac size and remodeling.
Change in Stroke Volume (SV) | Baseline, 6 Months Post-treatment
  Measured by CMR as the difference between LVEDV and LVESV.

SECONDARY OUTCOMES:
Total Clinical Effective Rate | 6 Months Post-treatment
  Assessed based on a composite of ECG improvement (including PVC burden reduction) and improvement in New York Heart Association (NYHA) functional class.
Change in Serum Heart-type Fatty Acid-Binding Protein (H-FABP) | Baseline, 6 Months Post-treatment
  Measured by ELISA as a biomarker for myocardial injury.
Change in Serum Soluble ST2 (sST2) | Baseline, 6 Months Post-treatment
  Measured by ELISA as a biomarker for myocardial fibrosis and inflammation.
Change in Serum Galectin-3 (Gal-3) | Baseline, 6 Months Post-treatment
  Measured by ELISA as a biomarker for myocardial fibrosis.
Change in Serum Tissue Inhibitor of Metalloproteinase-1 (TIMP-1) | Baseline, 6 Months Post-treatment
  Measured by double-antibody sandwich method as a biomarker related to extracellular matrix regulation.
Incidence of Adverse Events | Through study completion, an average of 6 months
  Number of participants experiencing any adverse events, including procedural complications, medication side effects, and arrhythmia recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Zhangjiakou City, Zhangjiakou, Hebei, China